CLINICAL TRIAL: NCT02338921
Title: Therapeutic Efficacy and Safety of Sitagliptin, Dapagliflozin and Lobeglitazone in Patients With Type 2 Diabetes Mellitus Inadequately Controlled on Glimepiride and Metformin.
Brief Title: Triple Combination Therapy in Type 2 Diabetic Patients Who Had Inadequate Glycemic Control With Combination Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Triple_3
Record Dates: First submitted 2015-01-11; First posted 2015-01-14 (Estimated); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Type 2 Diabetes
Keywords: triple combination therapy; sitagliptin; dapagliflozin; lobeglitazone
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; dapagliflozin; lobeglitazone; glimepiride; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Glimepirde, Metformin, Sitagliptin (Active Comparator): Dipeptidyl peptidase-4 (DPP4) inhibitor
  Sitagliptin
  Interventions: Drug: Sitagliptin; Drug: Glimepirde; Drug: Metformin
- Glimepirde, Metformin, Dapagliflozin (Active Comparator): Sodium-glucose cotransporter 2 (SGLT2) inhibitors
  Dapagliflozin
  Interventions: Drug: Dapagliflozin; Drug: Glimepirde; Drug: Metformin
- Glimepirde, Metformin, Lobeglitazone (Active Comparator): Peroxisome proliferator-activated receptor gamma agonist
  Lobeglitazone
  Interventions: Drug: Lobeglitazone; Drug: Glimepirde; Drug: Metformin

INTERVENTIONS:
Drug: Sitagliptin — 100mg qd per oral during 24months
  compared with other treatment groups
  Other Names: Januvia
  Arms: Glimepirde, Metformin, Sitagliptin
Drug: Dapagliflozin — 10mg qd per oral during 24months
  compared with other treatment groups
  Other Names: Forxiga
  Arms: Glimepirde, Metformin, Dapagliflozin
Drug: Lobeglitazone — 0.5mg qd per oral during 24months
  compared with other treatment groups
  Other Names: Duvie
  Arms: Glimepirde, Metformin, Lobeglitazone
Drug: Glimepirde
  Other Names: Amaryl
Drug: Metformin

SUMMARY:
To assess the efficacy of treatment with sitagliptin or dapagliflozin or lobeglitazone in type 2 diabetes mellitus patients, who had inadequate glycemic control even though use of two drug combination therapy with glimepiride and metformin.

DETAILED DESCRIPTION:
Dual combination therapy with metformin and sulphonylurea is the most commonly used combination regimen to treat patients with type 2 diabetes. But, treatment with the dual combination therapy is often unsuccessful at achieving glycaemic control in patients with type 2 diabetes.

Recently, various oral hypoglycemic agents were developed including dipeptidyl peptidase (DPP)-IV inhibitor, sodium-glucose cotransporter 2 (SGLT2) inhibitor and new peroxisome proliferator-activated receptors (PPARs) agonists.

But, there have been few studies about the glucose lowering effect of these drugs in Type 2 diabetes patients on the dual combination therapy with a sulfonylurea agent and metformin.

Hence, the researchers plan to investigate the efficacy and safety of these drugs in combination with a sulfonylurea agent and metformin in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* 20 ≤ Age < 80 years
* HbA1c ≥ 7 %
* combination therapy with glimepiride and metformin over 2 months.
* dosage of glimepiride : 1-8mg/day
* dosage of metformin : 500-2550mg/day

Exclusion Criteria:

* Type 1 diabetes, gestational diabetes, or secondary forms of diabetes
* Contraindication to sitagliptin or dapagliflozin or lobeglitazone
* Pregnant or breast feeding women
* Medication which affect glycemic control (ex. steroid)
* Disease which affect efficacy and safety of drugs
* Any major illness (Liver disease, Renal failure, Heart disease, Cancer, etc)
* Not appropriate for oral antidiabetic agent

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Glycemic target goal achievement rate | 24 months
  HbA1c< 7.0% without hypoglycemia

SECONDARY OUTCOMES:
Beta-cell function | 6 and 24 months
  Beta-cell function
insulin resistance | 6 and 24 months
  insulin resistance
Fasting blood sugar (FBS) and Post Prandial 2 hour blood glucose (PP2) | 3,6,9,12,16,20 and 24months
  Fasting blood sugar (FBS) and Post Prandial 2 hour blood glucose (PP2)
Lipid profile | 3,6,9,12,16,20 and 24months
  Lipid profile
Body fat | 6,12 and 24 months
  Body fat
urine microalbumin to creatinine ratio | 6,12 and 24 months
  urine microalbumin to creatinine ratio
Change of HbA1c | 3,6,9,12,16,20 and 24months
  Change of HbA1c
Glycemic target goal achievement rate | 12 months
  HbA1c< 7.0% without hypoglycemia

OTHER OUTCOMES:
hypoglycemia | 3,6,9,12,16,20 and 24months
  hypoglycemia
body weight change | 6 and 24 months
  body weight change

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, MD, PHD, Principal Investigator — SNUBH
Locations (1):
- Soo Lim, Seongnam-si, Gyeonggi-do, South Korea